CLINICAL TRIAL: NCT07247903
Title: The Effect of Virtual Reality-Based Education on Preoperative Surgical Fear, Postoperative Pain and Patient Satisfaction in Patients Undergoing Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: The Impact of Patient Education Delivered Through Virtual Reality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, KAHacıosmanoğlu, PhD student, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AnkaraYBU-HEM-KAH-01
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Knee Arthroplasty
Keywords: virtual reality; pain; surgical fear; patient satisfaction; knee arthroplasty
MeSH Terms: conditions — Pain; Patient Satisfaction | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomization Patients who meet the inclusion criteria for the study will be numbered sequentially starting from 1 and assigned using the block randomization method. These numbers will be randomly and equally divided into two groups-the control group and the experimental group-using a computer-assisted program.
Who Masked: Outcomes Assessor
Masking Description: Blinding of the Study and Prevention of Bias Assignment to control and experimental groups will be performed by an independent statistician to prevent bias and ensure confidentiality, and a blinding technique will be applied. Thus, selection bias will be controlled by random assignment and concealment of randomization. Since the intervention will be administered by the researcher, double-blinding will not be possible, but the data will be coded as 'A' and 'B' by the researcher and transferred to the computer. Furthermore, to prevent bias, the analysis of the coded data will be performed by an independent statistician outside the research team. The study protocol will follow the SPIRIT guidelines, and the reporting of the research will be conducted according to the Consolidated Standards of Reporting Trials (CONSORT) 2017 checklist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients who agree to participate in the study will be asked to complete a patient characteristics form. Patients in the control group will not receive any specific education from the researcher during the preoperative period. These patients will receive the clinic's routine patient education prior to surgery. After consulting with the nurses who provided the routine patient education at the clinic, the surgical fear scale will be administered. Upon arrival at the clinic after surgery, pain assessment will be performed using the VAS at 15 and 30 minutes, 1, 2, 4, 8, 12, and 24 hours. Since the data collection process for our study ends at 24 hours, the patient satisfaction scale will be completed at that time. Data collection is expected to take a total of 15-20 minutes.
- Experimental (Other): The researcher will provide patients with information about the virtual reality headset. The virtual reality headset will be disinfected before use for each patient. Patients in the experimental group will receive patient education using an animation-based video method with the virtual reality (VR) headset one day before the surgery. The training will be provided in a quiet, calm environment where the training will not be interrupted, in their own rooms for patients staying in single rooms, and in the nurse's room for patients staying in rooms with 2 or more beds. Patient education will be provided using the animation-based video method, and after answering the patient's questions, the surgical fear scale will be applied. Upon arrival at the clinic after surgery, pain assessment will be performed using the VAS at 15 and 30 minutes, 1, 2, 4, 8, 12, and 24 hours. Since the data collection process for our study ends at 24 hours, the patient satisfaction scale will be completed at that ti
  Interventions: Other: education

INTERVENTIONS:
Other: education — The preparation of patient education using animation-based video methods will first involve the researcher developing a scenario based on the literature, covering the preoperative preparation process, deep breathing and coughing exercises, Respiratory Exercise Device use, pain management, potential postoperative complications, wound care, mobilization, and the rehabilitation process. After the educational content and its suitability are reviewed and approved by 5 experts and its content validity is established, it will be forwarded to a graphic design expert for the preparation of the animation. Regular feedback will be obtained throughout the video preparation process, and the work will be closely monitored. The voiceover for the animation video will be done by the researcher.
  Arms: Experimental

SUMMARY:
Objective: A randomized controlled trial was designed to determine the effect of virtual reality-based education provided to patients undergoing knee arthroplasty on preoperative surgical fear, postoperative pain, and patient satisfaction.

Materials and Methods: The study was designed as a randomized controlled experimental study, with the group receiving animation-based patient education via virtual reality goggles serving as the experimental group and the group receiving routine patient education at the clinic serving as the control group. Research data will be collected using a patient characteristics form prepared by the researcher based on a literature review, a surgical fear scale, a visual analog scale, and a patient education satisfaction scale. Virtual reality glasses will be used as the application tool in the study.

DETAILED DESCRIPTION:
Type of Study The study was designed as a randomized controlled trial to determine the effect of virtual reality training provided to patients undergoing knee arthroplasty on preoperative surgical fear, postoperative pain and patient satisfaction.

Location and General Characteristics of the Study The study will be conducted at the Orthopedics and Traumatology Clinic of Ankara Gazi University Health Research and Application Center with patients who meet the study criteria.

Study Population and Sample The study population will consist of patients hospitalized at the Orthopedics and Traumatology Clinic of Ankara Gazi University Health Research and Application Center. Within this scope, the sample of the study will consist of patients selected by randomization from among individuals who will undergo knee arthroplasty surgery, in accordance with the inclusion and exclusion criteria of the study.

Blinding and Prevention of Bias in the Study Assignment to the control and experimental groups will be performed by an independent statistician to prevent bias and ensure confidentiality, and a blind technique will be applied. Thus, selection bias will be controlled by random assignment and concealment of randomization. Since the intervention will be administered by the researcher, double-blinding will not be possible, but the data will be transferred to the computer by the researcher and coded as 'A' and 'B'. Additionally, to prevent bias, the analysis of coded data will be conducted by an independent statistician outside the research team. The study protocol will follow the SPIRIT guidelines, and the research will be reported according to the Consolidated Standards of Reporting Trials (CONSORT) 2017 checklist.

Data Collection Tools Research data will be collected using a patient characteristics form prepared by the researcher based on a literature review, a surgical fear scale, a visual analog scale (VAS-pain), and a patient education satisfaction scale. Virtual reality glasses will be used as the application tool in the study.

Data Collection In order to conduct the research, after obtaining approval from the Ethics Committee of Ankara Yildirim Beyazit University and institutional permission from the Ankara Gazi University Health Research and Application Center, the researcher will explain the purpose of the study to the patients in the experimental and control groups and obtain an 'Informed Consent Form' from them before starting the application. The forms to be administered to patients will be completed by the researcher through face-to-face interviews.

Content of the Animation-Based Patient Education Provided To prepare patient education using animation-based video methods, the researcher will first prepare a scenario based on literature, covering the surgical preparation process, deep breathing and coughing exercises, Respiratory Exercise Device use, pain management, possible postoperative complications, wound care, mobilization, and the rehabilitation process. After the educational content and its suitability are reviewed and approved by 5 experts and its validity is confirmed, it will be sent to a graphic design expert for the preparation of the animation. Regular feedback will be obtained throughout the video preparation process, and the work will be closely monitored. The researcher will provide the voiceover for the animated video.

Research Plan A preliminary study group will be formed with patients who meet the research criteria and agree to participate in the study. After obtaining an 'Informed Consent Form' from the patients, the patient identification form will be completed. One day before surgery, patient education will be provided using an animation-based video method with virtual reality (VR) glasses. After receiving patient education and having their questions answered, the surgical fear scale will be applied. Upon arrival at the clinic after surgery, pain assessment will be performed using the VAS at 15 and 30 minutes, 1, 2, 4, 8, 12, and 24 hours. Since the data collection process for our study ends at 24 hours, the patient satisfaction scale will be completed at that time.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older,
* Agree to participate in volunteer work,
* Have no communication problems in terms of vision, hearing, and perception,
* Be able to read, speak, and understand Turkish,
* Have no fear of enclosed spaces.

Exclusion Criteria:

* Bilateral Total Knee Arthroplasty.
* Admission to the clinic on the day of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Fear Scale | one day before the surgery
  It is used to determine the fear levels of patients undergoing elective surgery. The scale consists of eight items on an 11-point Likert scale and is scored from zero to ten. The scale consists of two subscales that measure fear related to the short- and long-term outcomes of surgery. Items 1-4 measure fear of the short-term outcomes of the surgical procedure, while items 5-8 measure fear of the long-term outcomes of the surgical procedure. These questions address fears related to the surgical operation, anesthesia, pain, side effects, deterioration of health as a result of the surgical operation, failure of the surgical operation, inability to fully recover after the surgical operation, and prolongation of the recovery process. The items on the scale are rated on a scale of "0: not afraid at all" to "10: very afraid." The highest possible score on the scale is eighty, and the lowest is zero.

SECONDARY OUTCOMES:
Visual Analog Scale-Pain | Upon arrival at the clinic after surgery, pain assessment will be performed using the VAS at 15 and 30 minutes, and at 1, 2, 4, 8, 12, and 24 hours.
  The scale was developed by Price and colleagues in 1983 to determine the intensity of pain. It consists of a vertical or horizontal line measuring 10 cm in length, marked with different numbers. These numbers represent 0 = no pain and 10 = the most severe pain. The patient is asked to mark the current intensity of their pain on the scale. The length of the distance from the point indicating no pain to the marked point shows the intensity of the patient's pain. It is an easy-to-use and understandable measure for assessing pain intensity. In assessing pain intensity, <3 indicates mild pain, 4-6 indicates moderate pain, and >6 indicates severe pain.

OTHER OUTCOMES:
Patient Education Satisfaction Scale | It will be performed 24 hours after surgery.
  The scale, developed by Ciftci and colleagues in 2022, measures patient satisfaction levels with the education provided by healthcare professionals. It consists of thirty items and a single sub-dimension. There are no reverse items in the scale, and it is a Likert-type scale. Items are expressed as strongly disagree (1), disagree (2), undecided (3), agree (4), and strongly agree (5), and are evaluated by calculating the total mean scores of the scale items. The lowest possible score on the scale is 30, and the highest possible score is 150. As the score increases, the level of satisfaction with patient education increases. The Cronbach's alpha value of the scale is 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra AYMELEK HACIOSMANOĞLU, Principal Investigator

IPD SHARING:
Plan to Share IPD: No
I don't want to share until the app is finished